CLINICAL TRIAL: NCT05120479
Title: Effects of Taping on the Proprioceptive System of Healthy Subjects
Brief Title: Effects of Taping on the Proprioceptive System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Colexio Oficial de Fisioterapeutas de Galicia (Unknown)
Responsible Party: Principal Investigator, Lorenzo Antonio Justo Cousino, PhD, Physical Therapist, PhD., University of Vigo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: University of Vigo
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Athletic Tape; Proprioception; Wrist Joint; Arthrometry, Articular; Muscle Strength Dynamometer
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Masking Description: The forearm that is being evaluated will be hidden by a medical curtain so that the participants do not know the tape application that is being carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): The intervention will be the application of a Kinesiotape (KT) strip on the anterior side of the forearm.
  The day of the intervention will proceed as follows:
  * Warm-up: The total warm-up time will be 5 minutes. After warm-up, a 1 minute rest will be carried out.
  * Skin cleansing with 96% alcohol.
  * Kinesiotape (KT): KT will be placed without any extra tension (in the scientific literature it is called "paper off tension").
  Interventions: Procedure: Kinesiotape
- Control arm (Sham Comparator): The intervention will be the application of a tape strip on the anterior side of the forearm. Sham tape appears to be kinesiotape but is an inelastic tape.
  The day of the intervention will proceed as follows:
  * Warm-up: The total warm-up time will be 5 minutes. After warm-up, a 1 minute rest will be carried out.
  * Skin cleansing with 96% alcohol.
  * Sham tape: exactly the same procedure is followed as experimental arm, but an adhesive inelastic tape is used. Material: Omnifix elastic (Laboratorios Hartmann S.A .; Spain).
  Interventions: Procedure: Sham tape

INTERVENTIONS:
Procedure: Kinesiotape — Kinesiotape (KT): KT will be placed without any extra tension (in the scientific literature it is called "paper off tension"). The measure determined in the measurement with a tape measure is cut. The anchor of the KT is placed on the medial epicondyle with the body segments in a neutral position (anchor length: 5 cm). Placement of the active zone of the bandage with the flexor muscles of the fingers in elongation. Origin-insertion placement. Distal anchor in neutral position. Material: Kinesiotape: Kinesiology Tape TEMTEX ® Beige (Towatek Korea Co .; South Korea).
  Other Names: Kinesiology tape; Athletic tape
  Arms: Experimental arm
Procedure: Sham tape — Sham tape: exactly the same procedure is followed as above, but an adhesive inelastic tape is used. Material: Omnifix elastic (Laboratorios Hartmann S.A .; Spain).
  Arms: Control arm

SUMMARY:
Kinesiotape (KT) is a widely used technique, although the scientific evidence on its effectiveness is limited and conflicting. KT has not yet been scientifically proven to have an effect on proprioception and a possible placebo effect of this technique cannot be ruled out. The main objective of this experimental study is to evaluate the effect of the application of KT in the anterior side of the forearm on the force sense and the positional sense compared to a placebo intervention in healthy subjects. A randomized, single-blind, crossover clinical trial will be carried out, where each subject will undergo three situations in their dominant forearm: no intervention, intervention using sham tape and intervention using KT. In the present design, in a randomized manner, all subjects go through the 3 conditions on different days: KT, sham tape, and no intervention. Measurements will be made before and after the intervention and proprioception will be measured using the variables of sense of force (with a dynamometer) and joint position (with a goniometer). The main intervention will be the application of a KT strip on the anterior face of the forearm and a sham tape of another material following the same procedure. The study population will be made up of healthy students from the university community of the Faculty of Physiotherapy of the University of Vigo.

The main objective of this experimental study is to evaluate the effect of the application of kinesiotape (KT) in the anterior side of the forearm on the force sense and the joint positional sense of the wrist compared to a placebo/sham intervention in healthy subjects.

Study hypothesis: the application of KT on the anterior side of the forearm produces better results in the force sense evaluated by a grip dynamometry and on the joint position sense of the wrist compared to a sham intervention or not intervention.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be members of the University of Vigo who participate voluntarily in the study.
* Participants must be healthy subjects (men and women) of legal age (>18 years).
* All subjects must sign the informed consent prior to experimentation.

Exclusion Criteria:

* Suffering from dermal disorders, fragile skin or allergy to adhesive tape.
* Excessive skin hair in the region to apply the tape.
* Have received a bandage on the upper limb (MMSS) in two weeks prior to the experimentation.
* History of orthopedic / traumatic alterations in upper limb (deformities, arthropathy, muscular injuries, fracture or tendinopathy), neurological disorders (central or peripheral), systemic disorders, circulatory disorders (edema, heart failure, thrombosis, kidney failure), hormonal disorders or surgery in upper limb in the last 6 months.
* Have done strength training in the MMSS in the 48 hours prior to the study.
* Limitation in the range of motion of the MMSS that may affect the grip strength.
* Consumption of alcoholic beverages or medications 24 hours prior to the experimentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Force sense | 30 minutes
  Evaluation: ability of a subject to reproduce a certain force. Grip force.
  * Measuring instrument: dynamometer (JAMAR Smart Hand Dynamometer, Patterson Medical Holdings, Inc.).
Joint position sense | 30 minutes
  Evaluation: ability of a subject to reproduce a certain position. Wrist position.
  - Measuring instrument: goniometer (Baseline Bubble Inclinometer- Fabrication Enterprises USA and Universal Plastic Goniometer- Saehan Rulong Goniometer).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo A Justo Cousiño, PhD, Principal Investigator — Physiotherapy Group (FS1)- Faculty of Physiotherapy. University of Vigo
Locations (1):
- University of Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson B, Bialocerkowski A. The Effects of Kinesiotape Applied to the Lateral Aspect of the Ankle: Relevance to Ankle Sprains--A Systematic Review. PLoS One. 2015 Jun 23;10(6):e0124214. doi: 10.1371/journal.pone.0124214. eCollection 2015. PMID 26103637
- [Background] Csapo R, Alegre LM. Effects of Kinesio((R)) taping on skeletal muscle strength-A meta-analysis of current evidence. J Sci Med Sport. 2015 Jul;18(4):450-6. doi: 10.1016/j.jsams.2014.06.014. Epub 2014 Jun 27. PMID 25027771
- [Background] Parreira Pdo C, Costa Lda C, Hespanhol LC Jr, Lopes AD, Costa LO. Current evidence does not support the use of Kinesio Taping in clinical practice: a systematic review. J Physiother. 2014 Mar;60(1):31-9. doi: 10.1016/j.jphys.2013.12.008. Epub 2014 Apr 24. PMID 24856938
- [Background] Drouin JL, McAlpine CT, Primak KA, Kissel J. The effects of kinesiotape on athletic-based performance outcomes in healthy, active individuals: a literature synthesis. J Can Chiropr Assoc. 2013 Dec;57(4):356-65. PMID 24302784
- [Background] Kalron A, Bar-Sela S. A systematic review of the effectiveness of Kinesio Taping--fact or fashion? Eur J Phys Rehabil Med. 2013 Oct;49(5):699-709. Epub 2013 Apr 5. PMID 23558699
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Riemann BL, Lephart SM. The Sensorimotor System, Part II: The Role of Proprioception in Motor Control and Functional Joint Stability. J Athl Train. 2002 Jan;37(1):80-4. PMID 16558671
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702
- [Background] Reneker JC, Latham L, McGlawn R, Reneker MR. Effectiveness of kinesiology tape on sports performance abilities in athletes: A systematic review. Phys Ther Sport. 2018 May;31:83-98. doi: 10.1016/j.ptsp.2017.10.001. Epub 2017 Oct 9. PMID 29248350
- [Background] Poon KY, Li SM, Roper MG, Wong MK, Wong O, Cheung RT. Kinesiology tape does not facilitate muscle performance: A deceptive controlled trial. Man Ther. 2015 Feb;20(1):130-3. doi: 10.1016/j.math.2014.07.013. Epub 2014 Aug 6. PMID 25150913
- [Background] Zhang S, Fu W, Pan J, Wang L, Xia R, Liu Y. Acute effects of Kinesio taping on muscle strength and fatigue in the forearm of tennis players. J Sci Med Sport. 2016 Jun;19(6):459-64. doi: 10.1016/j.jsams.2015.07.012. Epub 2015 Jul 17. PMID 26229044
- [Background] Roijezon U, Clark NC, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 1: Basic science and principles of assessment and clinical interventions. Man Ther. 2015 Jun;20(3):368-77. doi: 10.1016/j.math.2015.01.008. Epub 2015 Jan 29. PMID 25703454
- [Background] Clark NC, Roijezon U, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 2: Clinical assessment and intervention. Man Ther. 2015 Jun;20(3):378-87. doi: 10.1016/j.math.2015.01.009. Epub 2015 Jan 29. PMID 25787919
- [Background] Kurt EE, Buyukturan O, Erdem HR, Tuncay F, Sezgin H. Short-term effects of kinesio tape on joint position sense, isokinetic measurements, and clinical parameters in patellofemoral pain syndrome. J Phys Ther Sci. 2016 Jul;28(7):2034-40. doi: 10.1589/jpts.28.2034. Epub 2016 Jul 29. PMID 27512259
- [Background] Han J, Waddington G, Adams R, Anson J, Liu Y. Assessing proprioception: A critical review of methods. J Sport Health Sci. 2016 Mar;5(1):80-90. doi: 10.1016/j.jshs.2014.10.004. Epub 2015 Feb 3. PMID 30356896
- [Background] Hagert E. Proprioception of the wrist joint: a review of current concepts and possible implications on the rehabilitation of the wrist. J Hand Ther. 2010 Jan-Mar;23(1):2-17. doi: 10.1016/j.jht.2009.09.008. Epub 2009 Dec 5. PMID 19963343